CLINICAL TRIAL: NCT03262831
Title: The Role of Mindful Movement in Women Receiving Adjuvant or Neoadjuvant Therapy for Breast Cancer
Brief Title: Mindful Movement in Women Receiving Adjuvant or Neoadjuvant Therapy for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Foundation for Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201708076
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer; Cancer of Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Yoga; Blood Specimen Collection; Weights and Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Yoga (Experimental): * Prior to start of treatment, a yoga therapist will work with each patient to develop a personalized yoga protocol using Gentle Hatha and Restorative Yoga
  * Each protocol will consist of 5-10 minutes of centering poses to invite focus and relaxation, then 15-20 minutes of seated and standing active poses, ending with 5-10 minutes of guided relaxation.
  * The personalized practice will be given to each participant and she will be asked to practice beginning at the start of neoadjuvant treatment at least 3 times a week (but preferably daily) at home for at least 30 minutes each time. Participants will continue their personalized yoga practice during the entirety of treatment. Each participant will be asked to journal when and for how long she practices at home and make any comments as to how the practice might have made her feel
  * During participation, weekly follow-up calls will be made by a member of the study team to each participant randomized to the yoga arm.
  Interventions: Other: Yoga; Procedure: Blood draw; Behavioral: FACT-G questionnaire; Procedure: Weight measurement; Behavioral: Recent Physical Activity Questionnaire; Behavioral: NHANES Food Questionnaire
- Arm 2: No Yoga (Active Comparator): -Patients in this arm will not receive a personalized yoga plan
  Interventions: Procedure: Blood draw; Behavioral: FACT-G questionnaire; Procedure: Weight measurement; Behavioral: Recent Physical Activity Questionnaire; Behavioral: NHANES Food Questionnaire

INTERVENTIONS:
Other: Yoga — The yoga practice, Gentle Hatha and Restorative Yoga, will be based on protocols that have been found to decease fatigue and weight gain by helping the participant gain insight in recognizing stress responses and ways to relax
  Arms: Arm 1: Yoga
Procedure: Blood draw — * Baseline and end of treatment
  * To evaluate change in inflammatory markers (CRP, IL-6, and TNF)
Behavioral: FACT-G questionnaire — * 7 statements that other people with breast cancer have said are important, the patient is to circle or mark one number per line to indicate the response as it applies in the last 7 days
  * Answers range from 0=not at all to 4=very much
Procedure: Weight measurement — -Weight will be taken at baseline, on day 1 of each cycle, and the end of treatment
Behavioral: Recent Physical Activity Questionnaire — -To assess physical activity, the RPAQ will be completed at baseline and at the end of treatment.
  Other Names: RPAQ
Behavioral: NHANES Food Questionnaire — -To assess diet, the NHANES Food Questionnaire will be completed at baseline and at the end of treatment.

SUMMARY:
The investigators hypothesize that a personalized yoga program with mindful movement implemented during breast cancer therapy will benefit women in multiple ways. The investigators predict that women participating in the program will experience less weight gain and fatigue and will have an improved quality of life compared to women not participating in the program. The investigators predict that this will be associated with decreased markers of inflammation. The investigators will also evaluate whether there is improved pathologic response rate compared to historical controls. This study will provide pilot data for a larger randomized controlled trial assessing whether program can provide long-term improvement in quality of life, weight maintenance, and the serum and tumor changes correlating with a reduced risk of recurrence and mortality.

ELIGIBILITY:
Eligibility Critera:

* Age ≥ 18.
* Female.
* Newly diagnosed with Stage I-III breast cancer.
* Scheduled to undergo neoadjuvant or adjuvant chemotherapy or neoadjuvant endocrine therapy.
* Not currently regularly practicing yoga (defined as at least once a month).
* Able to read and understand English
* Able to understand and willing to sign an IRB-approved written informed consent document

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Feasibility of enrolling patients to larger randomized controlled trial using yoga and mindful movement as measured the number of eligible patients enrolled | Completion of study enrollment (estimated to be 6 months)
  -Feasibility is defined as the ability to enroll 60% of eligible patients
Feasibility of conducting a larger randomized trial using yoga and mindful movement | Completion of study enrollment (estimated to be 6 months)
  -Feasibility is defined as the ability to have an 80% completion rate of the intervention
Efficacy of yoga exercise as measured by weight change from baseline to completion | Completion of treatment (estimated to be 6 months)

SECONDARY OUTCOMES:
Effect of yoga exercise as measured by rate of pathologic response (partial and complete) (neoadjuvant subset only) | Completion of treatment (estimated to be 6 months)
Effect of yoga exercise as measured by inflammatory markers | Completion of treatment (estimated to be 6 months)
Effect of yoga exercise as measured by fatigue index | Completion of treatment (estimated to be 6 months)
  -Fatigue index will be measured by FACT-G questionnaire
Effect of yoga exercise as measured by quality of life | Completion of treatment (estimated to be 6 months)
  -Quality of life will be measured by FACT-G questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay L Peterson, M.D., MSCR, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Greaney SK, Amin N, Prudner BC, Compernolle M, Sandell LJ, Tebb SC, Weilbaecher KN, Abeln P, Luo J, Tao Y, Hirbe AC, Peterson LL. Yoga Therapy During Chemotherapy for Early-Stage and Locally Advanced Breast Cancer. Integr Cancer Ther. 2022 Jan-Dec;21:15347354221137285. doi: 10.1177/15347354221137285. PMID 36412916
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu